CLINICAL TRIAL: NCT03966768
Title: DuraMesh Laparotomy Closure Following Trauma and Emergency Surgery
Brief Title: DuraMesh Laparotomy Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Mutual decision Walter Reed/U Maryland and Mesh Suture Inc.
Sponsor: Mesh Suture Inc. (Industry)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Laparotomy; Suture; Complications, Mechanical; Hernia Incisional
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Duramesh suturable mesh for laparotomy closure (Experimental): Patients undergoing a midline laparotomy for trauma or emergency surgery will be closed with Duramesh suturable mesh.
  Interventions: Device: Duramesh suturable mesh for laparotomy closure
- Conventional suture closure for laparotomy closure (Experimental): Patients randomized to conventional laparotomy closure will be closed using size 1 slowly-absorbing polydiaxonone (PDS) single strand or looped suture, based on surgeon preference.
  Interventions: Device: Conventional suture for laparotomy closure
- Open abdomen group closed in delayed fashion with Duramesh (Experimental): Patients undergoing delayed primary closure of an open abdomen will also be studied. 20 study patients undergoing delayed primary closure of an open abdomen will be closed with Number 1 or Number 2 Duramesh
  Interventions: Device: Duramesh suturable mesh for laparotomy closure

INTERVENTIONS:
Device: Duramesh suturable mesh for laparotomy closure — Patients undergoing laparotomy will be closed with Duramesh suturable mesh
  Arms: Duramesh suturable mesh for laparotomy closure; Open abdomen group closed in delayed fashion with Duramesh
Device: Conventional suture for laparotomy closure — Patients undergoing laparotomy will be closed with conventional polydiaxonone suture
  Arms: Conventional suture closure for laparotomy closure

SUMMARY:
This is a multisite randomized control proof-of-concept trial to evaluate the safety of Duramesh laparotomy closure in the trauma and emergency laparotomy setting. The study will be performed at University of Maryland Shock Trauma Center and Walter Reed National Military Medical Center. One hundred (100) patients will be randomized (2:1) to Duramesh laparotomy closure versus conventional suture closure.

After the patient has been confirmed to be a candidate for the trial, randomization will be performed in the operating room upon completion of the index abdominal procedure. Duramesh will be provided for patients assigned to the Duramesh treatment arm. Patients will be followed for 1 year following laparotomy closure at follow-up intervals of 1 month, 3 months, 6 months, and 12 months.

DETAILED DESCRIPTION:
Primary Laparotomy Closure Treatment 1) Study Group - Duramesh Laparotomy Closure (DLC) Treatment 2) Control Group - Conventional Suture Closure (CSC)

Patients undergoing a midline laparotomy for trauma or emergency surgery will have their abdominal wall laparotomy incision closed with size 0 Duramesh suturable mesh. Patients randomized to conventional laparotomy closure will be closed using size

1 slowly-absorbing (PDS) single strand or looped suture, based on surgeon preference.

While it would be preferable to identify a single conventional suture to serve as the control group, polling of potential participating surgeons demonstrated a preference for both single strand and looped sutures to be available for use in the conventional suture closure group. Both Duramesh and conventional sutures will be placed using a standardized closure technique that incorporates 1cm wide bites and 1cm spacing, as this is the established technique for trauma and emergency laparotomy closure at both participating institutions. An effort to quantify suture to wound length ratio will be made in an effort to confirm standardization of closure technique between groups. The small-bites surgical closure technique popular in Europe has not been adopted by trauma and emergency surgeons at either institution given concerns related to early dehiscence and the inability to extrapolate the STITCH trial data to a US trauma population. The surgeons at both institutions do not believe it acceptable to generalize the European trial with a mean BMI of 24 to the United States population, nor do they believe it wise to close the abdominal wall with a 2-0 polydioxanone suture, as this technique trended towards a higher rate of acute fascial dehiscence (burst abdomen).

All patients will be assessed for post-operative complications ( i . e . , infection, seroma, hematoma), a t 1 , 3 , 6 , and 12 months p o s t o p e r a t i v e l y . Patient will also be assessed for incisional hernia formation at the same post-operative time points (1, 3, 6, 12 months). Hernia outcomes will be based on physical examination, with ultrasound used for any uncertainties. While surveillance imaging has been shown to be more sensitive for hernia detection, the primary purpose of this study is to compare the safety profile of Duramesh laparotomy closure to standard closure technique. Surveillance imaging for hernia identification is not a part of standard clinical practice at the participating study sites. The rate of clinically relevant hernias found on physical exam will be used to inform future efficacy studies, where routine surveillance imaging will be incorporated into the study design.

In addition to the patients undergoing primary laparotomy closure following an open trauma or emergency abdominal surgery, an additional subset of 20 patients undergoing delayed primary closure of an open abdomen will also be studied. These patients represent a particularly challenging clinical problem, for which there is no standard approach to repair. All 20 study patients undergoing delayed primary closure of an open abdomen will be closed with #1 or #2 Duramesh and followed according to the same post-operative protocol as those undergoing primary laparotomy closure. This subgroup is too small for randomization to provide useful data for comparison, and thus will be used to provide only a descriptive analysis of this early experience with delayed Duramesh closure of the open abdomen. The safety of Duramesh closure in this patient population can be extrapolated from the previously referenced experience of mesh strip closures in contaminated incisional hernias.

ELIGIBILITY:
Inclusion Criteria:

* Midline laparotomy greater than 5 cm in length
* Urgent or emergent surgery following trauma
* Urgent or emergent surgery for diverticulitis
* Large or small bowel obstruction, acute abdomen, or intra-abdominal hemorrhage.
* Open abdomen after midline laparotomy.

Exclusion Criteria:

* Prior hernia repair or existing abdominal mesh
* Metastatic cancer
* Pregnancy
* Immunosuppression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 1 month
  Superficial or deep infection of the surgical site
Surgical site infection | 3 months
  Superficial or deep infection of the surgical site
Surgical site infection | 6 months
  Superficial or deep infection of the surgical site
Surgical site infection | 12 months
  Superficial or deep infection of the surgical site

SECONDARY OUTCOMES:
Surgical site occurrence | 1 month
  Any complication related to the surgical site, including hematoma, seroma, dehiscence, fistula, small bowel obstruction, exposed suture, return to the operating room, readmission, or mortality
Surgical site occurrence | 3 months
  Any complication related to the surgical site, including hematoma, seroma, dehiscence, fistula, small bowel obstruction, exposed suture, return to the operating room, readmission, or mortality
Surgical site occurrence | 6 months
  Any complication related to the surgical site, including hematoma, seroma, dehiscence, fistula, small bowel obstruction, exposed suture, return to the operating room, readmission, or mortality
Surgical site occurrence | 12 months
  Any complication related to the surgical site, including hematoma, seroma, dehiscence, fistula, small bowel obstruction, exposed suture, return to the operating room, readmission, or mortality
Intraoperative and hospitalization endpoints | Within 30 days
  Details regarding abdominal wall closure
Intraoperative and hospitalization endpoints | Within 30 days
  Length of hospital stay
Intraoperative and hospitalization endpoints | Within 30 days
  Length of the laparotomy incision and length of suture remnant
Intraoperative and hospitalization endpoints | Within 30 days
  Size of Duramesh used
Hernia formation | anytime within 12 months
  Clinical development of an incisional hernia
Patient reported outcomes | 3 months
  NRS pain scale
Patient reported outcomes | 6 months
  NRS pain scale
Patient reported outcomes | 6 months
  HerQles
Patient reported outcomes | 6 months
  SF-36
Patient reported outcomes | 12 months
  HerQles
Patient reported outcomes | 12 months
  SF-36
Patient reported outcomes | 12 months
  NRS pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Souza, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR); Thomas Scalea, MD, Study Director — U Maryland Shock Trauma

IPD SHARING:
Plan to Share IPD: No
As per the sponsor wishes

REFERENCES:
- [Background] Dumanian GA, Lanier ST, Souza JM, Young MW, Mlodinow AS, Boller AM, Mueller KH, Halverson AL, McGee MF, Stulberg JJ. Mesh sutured repairs of contaminated incisional hernias. Am J Surg. 2018 Aug;216(2):267-273. doi: 10.1016/j.amjsurg.2017.10.025. Epub 2017 Oct 25. PMID 29108644
- [Background] Lanier ST, Dumanian GA, Jordan SW, Miller KR, Ali NA, Stock SR. Mesh Sutured Repairs of Abdominal Wall Defects. Plast Reconstr Surg Glob Open. 2016 Sep 28;4(9):e1060. doi: 10.1097/GOX.0000000000001060. eCollection 2016 Sep. PMID 27757361
- [Background] Dumanian GA, Tulaimat A, Dumanian ZP. Experimental study of the characteristics of a novel mesh suture. Br J Surg. 2015 Sep;102(10):1285-92. doi: 10.1002/bjs.9853. Epub 2015 Jul 8. PMID 26154703
- [Background] Souza JM, Dumanian ZP, Gurjala AN, Dumanian GA. In vivo evaluation of a novel mesh suture design for abdominal wall closure. Plast Reconstr Surg. 2015 Feb;135(2):322e-330e. doi: 10.1097/PRS.0000000000000910. PMID 25626817